CLINICAL TRIAL: NCT02925143
Title: Improving Neuromuscular Monitoring and Reducing Residual Neuromuscular Blockade Via E-learning - a Multicenter Interrupted Time Series Study (INVERT Study)
Brief Title: Improving Neuromuscular Monitoring and Reducing Residual Neuromuscular Blockade Via E-learning
Acronym: INVERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jakob Louis Thomsen, MD, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: JLT-NM5
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Neuromuscular Blockade
Keywords: Residual nerve blockade; Neuromuscular monitoring; Residual curarization; Neuromuscular blocking agents; E-learning; Web based learning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- E-learning course (Experimental)
  Interventions: Other: E-learning course in neuromuscular monitoring

INTERVENTIONS:
Other: E-learning course in neuromuscular monitoring — An e-learning course designed to assess the challenges and common problems experienced by anesthetists when monitoring the neuromuscular blockade during general anesthesia.

SUMMARY:
To assess the impact of an e-learning course in neuromuscular monitoring on the frequency of application of objective neuromuscular monitoring for assessment of depth of neuromuscular blockade in general anaesthesia and secondarily on the incidence of residual neuromuscular blockade after anesthesia.

We will collect data prospectively from 6 Danish anaesthesia departments from the time of intervention, using data from the Anaesthesia Information Management System (AIMS). Baseline data is obtained from another study based on the same data extraction procedure (NCT02914119).

ELIGIBILITY:
Inclusion Departments We will include the 6 largest anaesthesia departments in the Zealand Region of Denmark.

Anaesthetists We will include the following anaesthesia personnel as anaesthetists: nurse anaesthetists in training, nurse anaesthetists, first year residents in anaesthesiology, residents in the last 4 years of training in anaesthesiology, and specialist consultants in anaesthesia.

Patients We will include and collect data from all patients undergoing general anaesthesia with neuromuscular blockade in each data collection period. Patients, who are eligible more than once, i.e. undergoing general anaesthesia on more than one occasion, will be included in the analyses with a case for every general anaesthetic received.

Exclusion criteria We will exclude personnel without clinical functions, i.e. administrative personnel.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6525 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob L Thomsen, MD, Principal Investigator — Sponsor principal investigator
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
Sharing of data not included in the permissions granted by authorities stated below

REFERENCES:
- [Derived] Thomsen JLD, Mathiesen O, Hagi-Pedersen D, Skovgaard LT, Ostergaard D, Gatke MR; INVERT collaborator group. Improving neuromuscular monitoring and reducing residual neuromuscular blockade via e-learning: A multicentre interrupted time-series study (INVERT study). Acta Anaesthesiol Scand. 2022 May;66(5):580-588. doi: 10.1111/aas.14038. Epub 2022 Feb 13. PMID 35122234
- [Derived] Thomsen JLD, Mathiesen O, Hagi-Pedersen D, Skovgaard LT, Ostergaard D, Engbaek J, Gatke MR. Improving Neuromuscular Monitoring and Reducing Residual Neuromuscular Blockade With E-Learning: Protocol for the Multicenter Interrupted Time Series INVERT Study. JMIR Res Protoc. 2017 Oct 6;6(10):e192. doi: 10.2196/resprot.7527. PMID 28986337

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-learning Course
Started | 6525
Participants Receiving Depolarizing Neuromuscular Blocking Agent (NMBA) (Succinylcholine) | 3099
Participants Receiving Non-depolarizing Neuromuscular Blocking Agent (NMBA) | 3426
Completed | 6525
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | E-learning Course
Number analyzed (Participants) | 6525
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3597
  Male | 2928
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 6525

OUTCOME MEASURES:

1. Primary Outcome: Application of Objective Neuromuscular Monitoring (Acceleromyography) in Cases Receiving a Depolarizing Neuromuscular Blocking Agent (NMBA) (Succinylcholine) (Yes/no)
Description: Number of Participants Who Received a Depolarizing Neuromuscular Blocking Agent (NMBA) (Succinylcholine) and was Monitored with Objective Neuromuscular Monitoring (Acceleromyography). Data on neuromuscular monitoring is automatically registered in the electronic patient chart when the equipment for acceleromyography is activated.
Time Frame: in the period from induction of anaesthesia to termination of anaesthesia, usually 2 hours
Population: Only patients who received a Depolarizing Neuromuscular Blocking Agent (NMBA) (Succinylcholine) are analyzed in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | E-learning Course
Number analyzed (Participants) | 3099
Participants | 1425

2. Primary Outcome: Application of Objective Neuromuscular Monitoring (Acceleromyography) in Cases Receiving a Non-depolarizing NMBA (Yes/no)
Description: Number of Participants Who Received a Non-depolarizing Neuromuscular Blocking Agent (NMBA) and was Monitored with Objective Neuromuscular Monitoring (Acceleromyography). Data on neuromuscular monitoring is automatically registered in the electronic patient chart when the equipment for acceleromyography is activated.
Time Frame: in the period from induction of anaesthesia to termination of anaesthesia, usually 2 hours
Population: Only patients receiving a non-depolarizing neuromuscular blocking agent are analyzed in this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | E-learning Course
Number analyzed (Participants) | 3426
Participants | 3172

3. Secondary Outcome: Last Recorded Train-of-four (TOF) Ratio Before Tracheal Extubation or Removal of Supraglottic Airway Device in Patients Receiving a Non-depolarizing NMBA
Description: The Train-of-four (TOF) ratio is the ratio of the fourth to the first muscle response after 4 stimuli at the ulnar nerve at the wrist at 2 Hz. The response is measured using acceleromyography. If the last measurement is performed before return of any muscle function, the ration can not be given.
Time Frame: in the period from induction of anaesthesia to termination of anaesthesia, usually 2 hours]
Population: Only patients receiving a non-depolarizing neuromuscular blocking agent, monitored with acceleromyography and with a valid TOF ratio in the last three measurements are included in this outcome.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | E-learning Course
Number analyzed (Participants) | 3027
ratio | 95.23 (29.57)

4. Secondary Outcome: Administration of Sugammadex in Cases Receiving a Non-depolarizing NMBA (Yes/no)
Description: If the total dose of sugammadex in the anaesthesia information management system is > 0, the outcome is "yes".
Time Frame: in the period from induction of anaesthesia to discharge from the post-anaesthesia care unit, usually 5 hours
Population: Only patients receiving a non-depolarizing neuromuscular blocking agent are analyzed in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | E-learning Course
Number analyzed (Participants) | 3426
Participants | 85

5. Secondary Outcome: Administration of Neostigmine in Cases Receiving a Non-depolarizing NMBA (Yes/no)
Description: If the total dose of neostigmine in the anaesthesia information management system is > 0, the outcome is "yes".
Time Frame: in the period from induction of anaesthesia to discharge from the post-anaesthesia care unit, usually 5 hours
Population: Only patients receiving a non-depolarizing neuromuscular blocking agent are analyzed in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | E-learning Course
Number analyzed (Participants) | 3426
Participants | 2047

6. Secondary Outcome: Administration of More Than One Reversal Agent in Cases Receiving a Non-depolarizing NMBA (Yes/no)
Description: If the total dose of neostigmine is bigger than (>) the first dose administered, the outcome is "yes".
Time Frame: in the period from induction of anaesthesia to discharge from the post-anaesthesia care unit, usually 5 hours
Population: Only patients receiving a non-depolarizing neuromuscular blocking agent are analyzed in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | E-learning Course
Number analyzed (Participants) | 3426
Participants | 213

7. Secondary Outcome: Time in Minutes From Tracheal Extubation or Removal of Supraglottic Airway Device to Discharge From Post-anaesthesia Care Unit in Cases Involving a Non-depolarizing NMBA
Time Frame: in the period from induction of anaesthesia to discharge from the post-anaesthesia care unit, usually 180 minutes
Population: Only patients receiving a non-depolarizing neuromuscular blocking agent with data on length-of-stay in the post-anaesthesia care unit are analyzed in this outcome.
Measure: Median (Full Range); unit: minutes
Arm/Group | E-learning Course
Number analyzed (Participants) | 2533
minutes | 100 [1 to 1431]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | E-learning Course
All-Cause Mortality (participants affected / at risk) | 0/6525
Serious Adverse Events (participants affected / at risk) | 0/6525
Other Adverse Events (participants affected / at risk) | 0/6525

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT02925143/Prot_SAP_000.pdf